CLINICAL TRIAL: NCT05770050
Title: Cardiac Changes Associated With Acute Cerebrovascular Stroke
Brief Title: Cardiac Changes Associated With Acute Cerebro-vascular Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Ali, Esraa Mohamed Ali, Assiut University
Other Study IDs: CVS and Cardiac changes
Record Dates: First submitted 2023-03-02; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Cardiovascular disease is regarded as main predisposing risk factor for cerebrovascular stroke.

Cardiac dysfunction can both worsen the pre existing cerebral damage and cause new brain injury Diseases of the heart and the brain are closely entangled. Vascular diseases of both organs share the same risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. above 18 years
2. patients presented with cerebrovascular stroke 3-patients diagnosed as cardiac patients and have cerebrovascular stroke

Exclusion Criteria:

1-Less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with acute cerebrovascular accident and have cardiac diseases are investigated by ECG, Echo, Troponin level to detect different cardiac abnormalities associated with cerebrovascular accident
Sampling Method: Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
ECG changes in cerebrovascular accident | 6 months
  ECG QT interval, T wave changes in. cerebrovascular accident
Echo changes in cerebrovascular accident | 6 months
  Echo chamber dilatation, valavular, ejection fraction changes in cerebrovascular accident